CLINICAL TRIAL: NCT06796504
Title: The SetPoint System as a Pro-Remyelination Therapy for Relapsing-Remitting Multiple Sclerosis: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPM-040
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Active stimulation for 1 minute once per day
  Interventions: Procedure: Procedure/Surgery: Implant Procedure; Drug: Disease-Modifying Therapies (DMTs); Device: Device: Active stimulation
- Control (Sham Comparator): Non-active stimulation for 1 minute once per day
  Interventions: Procedure: Procedure/Surgery: Implant Procedure; Drug: Disease-Modifying Therapies (DMTs); Device: Device: Non-active stimulation

INTERVENTIONS:
Procedure: Procedure/Surgery: Implant Procedure — The SetPoint System (study device)contains a miniaturized stimulator (implnat) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). All eligible subjects will undergo the surgery under general anesthesia in outpatient settings.
Drug: Disease-Modifying Therapies (DMTs) — All subjects will continue treatment with standard of care disease-modifying therapies for he duration of the study.
Device: Device: Active stimulation — Active stimulation for 1 minute once per day
  Arms: Treatment
Device: Device: Non-active stimulation — Non-active stimulation for 1 minute once per day
  Arms: Control

SUMMARY:
The MS pilot study will assess the safety and investigate the remyelinating effects of the SetPoint System (study device) in adult patients with patients diagnosed with relapsing-remitting multiple sclerosis (RRMS). The SetPoint System is intended for adjunctive use with standard of care therapy for RRMS. The study device contains a miniaturized stimulator (implant) that is surgically placed under general anesthesia on the vagus nerve through a small incision on the left side of the neck (implant procedure). The study will enroll up to 60 participants at up to 10 sites. All eligible participants will undergo the implant procedure. Two-thirds of the participants will receive active stimulation (treatment) and the one-third will receive non-active stimulation (control). Following treatment evaluations at Week 48, there will be a one-way crossover of control subjects to active stimulation and a 48-week open-label follow-up with all subjects (treatment and control) receiving active stimulation to evaluate long-term safety.

DETAILED DESCRIPTION:
The MS pilot study is a 2:1 randomized, double-blind, sham-controlled, multi-center pivotal study enrolling up to 60 subjects at up to 10 study centers across the U.S. The study will assess the safety and investigate the remyelinating effects of the SetPoint System (study device) in adult patients with patients diagnosed with relapsing-remitting multiple sclerosis (RRMS). The SetPoint System is intended for adjunctive use with standard of care therapy for RRMS. The study device contains a miniaturized stimulator (implant) that is surgically implanted inside the left side of the neck on the vagus nerve (implant procedure). The implant delivers a small amount of electricity (stimulation) to the nerve. All eligible subjects will undergo the surgery under general anesthesia. Two-thirds of the subjects will receive active stimulation (the treatment group) and the other one-third will receive non-active stimulation (the control group). Stimulation will be delivered for 1 min once per day for 48 weeks. Following treatment evaluations at Week 48, there will be a one-way crossover of control subjects to active stimulation and a 48-week open-label follow-up with all subjects (treatment and control) receiving active stimulation to evaluate long-term safety. Blinding will be maintained for each individual participant until that participant has completed their Week 48 assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-50 years at informed consent.
* Diagnosis of RRMS by revised 2017 McDonald criteria.
* Latency delay >118 milliseconds on baseline full-field transient pattern reversal visual evoked potential (VEP) in at least one eye. Both eyes can be included if they meet all inclusion criteria.
* Peri-papillary retinal nerve fiber layer (pRNFL) > 70 microns on Optical Coherence Topography (OCT) in the VEP-qualifying eye (sufficient axons).
* Best corrected high-contrast (HCVA) better than 20/200 Snellen equivalent or letter score of 35
* Best corrected low-contrast letter acuity (LCLA) by Sloan chart (2.5% black on white) of no better than 40 letters in the VEP-qualifying eye (Snellen equivalent of 20/40). (Best corrected LCLA must be worse than best corrected HCVA.)
* Absence of clinical relapse for at least 12 months prior to informed consent
* No new lesions or increase in existing lesion volume on most recent clinic brain MRI (must be within 1 year of consent)
* Taking a stable regimen of disease-modifying therapy (DMT) prior to informed consent. If intermediate-potency DMT, the DMT must have been started and maintained for at least two years prior to consent. If high-potency DMT, the DMT must have been started and maintained at least one year prior to consent.
* Score of 2.5 to 6.0 by Expanded Disability Status Scale (EDSS) at baseline, with at least of 2 on the functional systems pyramidal function.

Exclusion Criteria:

* Confounding ophthalmologic disease or impairments/conditions that could interfere with visual testing (e.g., cataracts, disc hemorrhage, macular star, cotton wool spots, macular degeneration, glaucoma, diabetic and/or hypertensive retinopathy, history of detached retina, etc.)
* Severe myopia defined as a refractive error of -6.00 diopters or more
* Concurrent neurological disorders, including known moderate or severe cervical myelopathy.
* Clinical optic neuritis within 6 months before screening.
* Documented optic neuritis in the qualifying eye greater than 5 years before screening.
* Steroid treatment for MS symptoms in the 30 days prior to consent
* Hypersensitivity/allergy to MRI contrast agents and/or unable to perform MRI (e.g., claustrophobia).
* Regular use of or dependency on nicotine products within the past year.
* Not a surgical candidate.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Informed consent through Week 96
  All adverse events from Screening through Week 96 (end of study) will be tabulated.

OTHER OUTCOMES:
Reduction in VEP latency | Baseline (Screening) through Week 48
  Change from baseline full-field VEP P100 latency at Week 48.
Change in lesion size as detected on MRI | Baseline (Screening) through Week 48
  New T2 and/or contrast enhancing lesions Change in T2 lesion volume Change in phase (paramagnetic) rim lesions (PRL) Difference in the occurrence and volume of slowly expanding lesions
Change in number of letters accurately read | Baseline (Screening) through Week 48
  Change from baseline in LCLA and HCVA at Week 48.
Change in the NEI-VFQ-25 score | Baseline (Screening) through Week 48
  Change from baseline in NEI-VFQ-25 at Week 48
Change in EDSS scores | Baseline (Screening) through Week 48
  Change from baseline in EDSS at Week 48
Change in Modified MSFC scores | Baseline (Screening) through Week 48
  Change from baseline in modified MSFC at Week 48 for both composite score and each individual assessment (25-foot timed walk, 9-hole peg, and Symbol Digit Modalities Test)
Change in MFIS score | Baseline (Screening) through Week 48
  Change from baseline in MFIS at Week 48
Change in magnetization transfer ratios (MTR) in brain lesions | Baseline (Screening) through Week 48
  MTR is a surrogate to detect remyelination of lesions in the brain.

IPD SHARING:
Plan to Share IPD: No